CLINICAL TRIAL: NCT06023186
Title: Coronary Flow Reserve in oHCM Patients Before and After 12 Months of Standard-of-care Mavacamten Treatment as Assessed by PET/CT
Brief Title: Effect of Mavacamten Treatment on Coronary Flow Reserve in oHCM
Acronym: MavaPET
Status: Recruiting | Type: Observational
Sponsor: Michael Ayers (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Michael Ayers, Assistant Professor, University of Virginia
Organization: University of Virginia (Other)
Other Study IDs: HSR220293
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Clinically stable, adult patients with obstructive hypertrophic cardiomyopathy, who meet mavacamten prescribing guidelines will be prescribed mavacamten by their treating physician.
  Interventions: Drug: mavacamten

INTERVENTIONS:
Drug: mavacamten — Study participants will receive mavacamten under the standard of care
  Other Names: Camzyos

SUMMARY:
The goal of this observational study is to measure the effect of mavacamten treatment on blood flow in the heart muscle (myocardium) in patients with obstructive hypertrophic cardiomyopathy. The main question it aims to answer is:

• Does mavacamten treatment improve blood flow in the heart muscle?

Participants will take mavacamten at the direction of their treating physician. Participants will complete 2 myocardial Positron Emission Tomography and Computed Tomography (PET-CT) scans. The first scan will be completed before participants start taking mavacamten. The scan will be repeated after 12 months of mavacamten treatment.

DETAILED DESCRIPTION:
This is a single-arm, before-and-after investigation of the effect of mavacamten therapy on myocardial blood flows in adult human subjects prescribed mavacamten for clinical standard of care for oHCM. We hypothesize that 12 months of mavacamten therapy will improve myocardial blood flows as assessed by PET/CT. The investigation will take place at a single site. Participants who consent will be prospectively enrolled once mavacamten therapy has been approved by their health insurance/payer. Enrolled participants will undergo myocardial PET/CT before starting mavacamten and after 12 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide written informed consent
2. Willingness and ability to comply with scheduled visits and study procedures
3. Male or female, aged 18-85 years
4. Diagnosed with obstructive hypertrophic cardiomyopathy according to presence of a left ventricular wall thickness of ≥15 mm that is otherwise unexplained by abnormal loading conditions (e.g., hypertension, valvular, congenital disease) or infiltrative cardiomyopathies. Unexplained left ventricular wall thickness of ≥13 mm is sufficient for diagnosis in relatives of individuals with hypertrophic cardiomyopathy or those who are genotype positive.
5. Has been prescribed mavacamten consistent with US Prescribing Information
6. Ability and intention to adhere to oral mavacamten therapy as prescribed by treating physician for the duration of study participation
7. For females of reproductive potential: negative pregnancy test at screening/baseline and 12 month visits.

Exclusion Criteria:

1. Pregnancy or lactation
2. Known hypersensitivity to components of mavacamten or regadenoson
3. Prior treatment with mavacamten or aficamten

11. Over weight limit for imaging gantry. 12. To minimize the risk of participants undergoing PET/CT with inadequate image quality, participants with left ventricular systolic dysfunction or lung disease will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable adult obstructive hypertrophic cardiomyopathy patients on background therapy who have been prescribed Camzyos (mavacamten) in accordance with the US Prescribing Information, but who have not yet started this medication.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial perfusion reserve after 12 months of mavacamten treatment. | 12 months
  Myocardial perfusion reserve is the ratio of global myocardial blood flow at stress versus rest.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No data on individual participants will be shared outside the University of Virginia.